CLINICAL TRIAL: NCT06432491
Title: Study to Explore How Core Temperature Reduction Influence Health
Brief Title: The Association Between Core Temperature and Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Collaborators: Shenzhen University General Hospital (Other); The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, John R. Speakman, Prof., Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KYLLHS-20240201A
Record Dates: First submitted 2024-05-01; First posted 2024-05-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Body Temperature Changes; Body Composition; Aging
Keywords: Body temperature; Body composition; Aging
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into intervention group and control group. Intervention group will drink 4℃ water while control group will drink 37℃ water for 6 months.
Who Masked: Participant, Investigator
Masking Description: All the participants will only get access to their own group and will not get access to other group members.
  The investigator who take charge of MRI test for participants' body composition will not have any idea about grouping.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4℃ water drinking group (Experimental): Volunteers will drink 500ml 4℃ water within 10 minutes at 9a.m., 12p.m., 15p.m., 18p.m. everyday for 6 months.
  Interventions: Behavioral: Drinking cold water
- 37℃ water drinking group (No Intervention): Volunteers will drink 500ml 37℃ water within 10 minutes at 9a.m., 12p.m., 15p.m., 18p.m. everyday for 6 months.

INTERVENTIONS:
Behavioral: Drinking cold water — Volunteers in the intervention group will be asked to drink up 500 ml 4℃ water within 10 minutes four times per day throughout the study.
  Arms: 4℃ water drinking group

SUMMARY:
The goal of this clinical trial is to learn if cold water drinking could promote body composition and further extend healthy lifespan in Chinese older adults. The main questions it aims to answer are:

1. Does cold water drinking lower the body fat percentage?
2. Will cold water drinking positively extend lifespan in a long-term Researchers will compare cold water intervention group to a control group (drinking 37℃ water instead) to see if cold water drinking works to promote health and slow down ageing process.

Participants will:

1. Drink 4℃ or 37℃ water 4 times (9a.m., 12p.m., 15p.m., 18p.m.) every day for 6 months.
2. Visit the institute and health checkup department for tests and checkup at baseline, the end of the 3rd month, and the end of 6th month.

DETAILED DESCRIPTION:
According to pilot study, we found 4℃ water could significantly reduce core body temperature. Thus, we aim to explore whether 4℃ water drinking could promote body composition and further help to extend lifespan.

Participants will be randomly divided into intervention (drinking 4℃ water at 9a.m., 12p.m., 15p.m., 18p.m.) and control group (drinking 37℃ water at 9a.m., 12p.m., 15p.m., 18p.m.) for 6-month intervention. Tests will be conducted in Shenzhen Institute of Advanced Technology, while checkup will be tested at Health Checkup Department of Shenzhen University General Hospital. Body composition will be tested by Magnetic Resonance Imaging (MRI), Dual-Energy X-Ray Absorptiometry (DEXA), and TANITA (bioelectrical method). In addition, we will test participants' waist and hip circumferences using 3D scanning. Besides, we will test core body temperature and brown adipose tissue.

Apart from above main outcomes, we will also test their physical activity, food intake, metabolic rate, glucose, IL-6, TNF-alpha, HDL, LDL, insulin level. Meanwhile, ageing biomarkers, namely Phenotypic Age, eye fundus image, facial changes, bone density, gut microbiota, GlycanAge, will also be measured.

The whole intervention period will last for 6 months. All the tests and checkup will be tested at baseline, the end of the third month and the endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 65 years old (including 50 and 65)
* No surgery in the past 6 months
* Healthy (No metabolic diseases, cardiovascular diseases, lung diseases (COPD, asthma, et al.), endocrine diseases and gastrointestinal diseases)
* Based in Shenzhen during the whole study period
* No significant change on body weight in the past 3 months

Exclusion Criteria:

* Those who need to take medication for a long term (including diet pills)
* On a diet
* Disabled
* Females who are trying to get pregnant, pregnant, or breastfeeding
* Presence of a metal implant in the body (e.g. pacemaker)
* Those with claustrophobia
* Those with blood phobia, pathological hypotension or hypertension
* Those who are in other intervention studies

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Value of core body temperature in centigrade assessed by e-Celsius | Twenty-four hours every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Volunteers will swallow an electronic capsule called e-Celsius (BodyCap, France) which will be activated before use. Four hours after swallowing, the e-Celsius will enter intestine and data collection will start. A device call e-Viewer (KIT EPERF CE-SW, France) will be used to connect the capsules and collect data.
Value of weight in kilogram assessed by Seca body weight scale | Five minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Volunteers will be asked to fast overnight and weight will be measured using a calibrated Seca body weight scale first thing in the morning on subjects wearing light clothes and no shoes.
Value of height in meters assessed by Seca 217 stadiometer | Five minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Measured by Seca 217 Stable Stadiometer. Volunteers should not wear shoes and socks. Stand on the stadiometer platform with back against the wall and feet together. Stand up as straight as possible with heels, back, shoulders, and head all touching the wall. Tuck in chin and look straight ahead.
Value of body mass index (BMI) calculated by weight and height | The calculation will cost two minutes every three months for the 6 months of the experiments.The calculation will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  BMI will be calculated based on weight and height according to the formula: BMI=Weight/Height^2
Body composition- volume of fat mass in cm^3 assessed by uMR 790 | Fifteen minutes every three months for the 6 months of the experiments.The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ). Volunteers should wear no metal jewelries or with metal implants. They should lie down on a movable table and be fasten by technologists. Volunteers should hold still during the test and perform a few small tasks, such as exhale, inhale, and hold breath following the broadcast.
Body composition-weight of fat free mass in gram assessed by Tanita MC-980 | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980). Demographic information of volunteers should be entered before test, including ID number, sex, age, height. When the signal showing the machine is ready, volunteers should stand on the scale without shoes, socks or any pieces which might influence weight. According to the instruction of display screen, volunteers need to hold the handle tightly.
Body composition-wegiht of fat mass in gram assessed by Horizon Wi | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Fat free mass will be measured by DEXA (Horizon Wi). Volunteers will be asked to lie on a special DEXA x-ray table. The technologist will help position your correctly and use positioning devices such as foam blocks to help hold the desired position. As the arm of the DEXA machine passes over the body, IT uses two different x-ray beams. The beams use very little radiation to keep the test safer, and help to distinguish bone from other tissues. The scanner translates the bone density measurement data into pictures and graphs. Bone is most easily seen in white, while the, fat and muscle tissue look like shadows in the background on the technologist's computer monitor.
Waist circumferences in centimeter assessed by TG2000-F | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Waist circumferences will be measured using a whole body laser scanner (TG2000-F). Volunteers should wear tight underwear during test and stand in front of the machine according to the stickers of instruction. Do some small movement according to instruction.
Hip circumferences in centimeter assessed by by TG2000-F | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Hip circumferences will be measured using a whole body laser scanner (TG2000-F). Volunteers should wear tight underwear during test and stand in front of the machine according to the stickers of instruction. Do some small movement according to instruction.
Brown adipose tissue-areas of temperature increase in cm^2 assessed by Fluke RSE600 | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  The infrared thermal imager (Fluke RSE600) will be used to measure brown adipose tissue around clavicle. Each subject was in a relaxed "steady-state" within a familiar environment. They were seated in an upright posture, with arms adducted and with head, neck, and shoulders unclothed, in the center of the study room, away from all heat-emitting objects and 1.0 m away from a thermal imaging camera fixed on a tripod at a set distance, 1 m, from the floor. This positioning ensured comfort as well as the optimum position for visualization of the supraclavicular BAT depots. 5 images were taken at 1-minute intervals before each thermal challenge and represented the control period. Each subject then placed 1hand into cool tap water (20℃).The increase in temperature in the thermal area in the supraclavicular region was further collected.

SECONDARY OUTCOMES:
Intensity of physical activity in three types (light, moderate, vigorous) assessed by GT3X | Seven days every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Physical activity of the volunteers will be recorded using accelerometer (GT3X) worn near the hip for a consecutive period of 7 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day where the wear time is less than 12 hours. For a valid measure the goal is to get 2 weekday and 2 weekend days. The acceleration of three axises will be collected and then calculated into the intensity of physical activity.
Weight of food intake in gram assessed by 24-hour Dietary Review Questionnaire | One day every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Food intake was monitored using the 24-hour Dietary Review questionnaire (a retrospective record of food intake (quantity and frequency) over the past 24 hours using a self-reported questionnaire).
Resting metabolic rate in kcal assessed by Cosmed | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Resting energy expenditure will be measured using indirect calorimetry via a respiratory hood system (Cosmed). The volunteer attends in the lab after an overnight fast. The person lies down on a flat bed and the hood is placed over their head. Metabolic rate (oxygen consumption and CO2 production) are monitored for 40 minutes. The last 10 minutes is used as the measurement. Calorimeters will be assessed with a turbine test to ensure accuracy of measurements. Validation via an alcohol burn will be performed monthly.
Concentration of glucose in mmol/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for glucose test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of IL-6 in ng/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for IL-6 test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of TNF-Alpha in ng/mL assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for TNF-Alpha test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of High-Density Lipoprotein (HDL) in mmol/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for HDL test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of Low-Density Lipoprotein (LDL) in mmol/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for LDL test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of triglyceride (TG) in mmol/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for TG test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of insulin in mU/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.

OTHER OUTCOMES:
Concentration of albumin in g/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of creatinine in umol/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of C-reactive protein in mg/dL assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Percentage of lymphocyte assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Volume of mean (red) cell assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Coefficient of variation of red blood cell size (red cell distribution width) assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Concentration of alkaline phosphatase in U/L assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Number of white blood cell (white blood cell count) in 1000 cells/uL assessed by clinical blood test | Fifteen minutes of blood test every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse for insulin test in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital.
Calculation of Phenotypic Age based on blood test | The calculation will cost 5 minutes. The calculation will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Venous blood sample will be collected by professional nurse in the morning after 12 hour fasting and be examined by Shenzhen University General Hospital. Index of albumin, creatinine, glucose, c-creative protein, lymphocyte percentage, mean corpuscular volume, red cell distribution width, alkaline phosphatase, white blood cell count will be examined and calculated into Phenotypic Age.
Bone density in g/cm^2 assessed by Horizon Wi | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Bone mass will be measured by DEXA (Horizon Wi). Volunteers will be asked to lie on a special DEXA x-ray table. The technologist will help position your correctly and use positioning devices such as foam blocks to help hold the desired position. As the arm of the DEXA machine passes over the body, IT uses two different x-ray beams. The beams use very little radiation to keep the test safer, and help to distinguish bone from other tissues. The scanner translates the bone density measurement data into pictures and graphs. Bone is most easily seen in white, while the, fat and muscle tissue look like shadows in the background on the technologist's computer monitor.
Eye fundus imaging assessed by Spectralis OCT | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Volunteers will go to the Health Management Center of Shenzhen University General Hospital, where professional doctors will use a photocoherence tomography scanner (Spectralis OCT) for fundus examination, and fundus imaging will be collected without invasiveness and harm. Volunteers need to sit comfortably in a chair and move their face close to the camera device. Technologist will show where to place forehead and chin. Nothing touches volunteers' eye during retinal imaging.
Picture of facial features assessed by Fluke RSE600 | Fifteen minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Facial features are captured using an infrared thermal imager (Fluke RSE600), which are then analyzed using artificial intelligence. When shooting, wait for the thermal imager to focus and press the shutter. During image acquisition, the frame should contain only one subject, whose face and head information are fully collected, and the area above the neck accounts for more than 35% of the thermal image captured. During the collection process, volunteers are reminded to look up at the camera, not to make expressions, not to wear glasses that cover their faces, masks, etc. In the event that the volunteer has bangs or long hair covering their face, the volunteer should be reminded to put on a headband and tie their hair back.
Muscle strength in kilogram assessed by Jamar Plus+ Digital Hand Dynamometer | Ten minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Muscle strength will be measure by Jamar Plus+ Digital Hand Dynamometer. Volunteers will comfortably arrange the instrument in his/her hand. Have volunteers squeeze with their maximum strength. The peak-hold needle will automatically record the highest force exerted.
Microbiome assessed by Illumina | Feces will be collected by volunteers themselves and send to the researchers. Feces will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  Abundance of gut microbiome will be from Metagenomic profiling of feces by Illumina. Volunteers will collect their feces by themselves using a specialized feces collection tubes. They need to submit the samples to the researcher within 30 minutes after collection or they need to first store in the freezer and then submit the sample when available.
Score of GlycanAge assessed by GlycanAge kit | Ten minutes every three months for the 6 months of the experiments. The data will be collected at baseline, the end of the 3rd month, and the end of the 6th month.
  The researcher will take a drop of blood from the volunteers' finger stick, use the kit to store the fingerstick blood, and then send it to the company for testing. Biological age score based on glycan biomarkers that indicate inflammation will be available in 3-5 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Chinese Academy of Sciences, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No